CLINICAL TRIAL: NCT07018609
Title: The Zen Den - Mitigating Burnout in Nursing and Associated Healthcare Staff
Brief Title: Mitigating Burnout in Nursing and Associated Healthcare Staff
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Eric Messner, Assistant Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study00026654
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Burn Out; Nurses
Keywords: Burnout; Nurses; Music Therapy
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zen Den (Active Comparator): Zen Den
  Interventions: Behavioral: Zen Den Experience
- Music Therapy (Active Comparator)
  Interventions: Behavioral: Music Therapy Experience

INTERVENTIONS:
Behavioral: Zen Den Experience — The Zen Den is a dedicated safe space for healthcare staff to decompress and recharge during shifts, addressing the growing issue of workplace stress. It has soft warm lighting, sound machines and aroma therapy, relaxing furnishings centered around a faux fireplace to create a stress-free environment.
  Arms: Zen Den
Behavioral: Music Therapy Experience — The music therapy experience will consist of either Music Minutes which have music therapists available on specific units and circulating amongst staff across flexible shift times. Intervention choices will include relaxation songs, motivation songs, music, mindfulness, breathing to music, dance-a-minute, and brief song rewrites. Notes for Resilience will be scheduled group sessions that follow a more structured format and are 30 to 60 minutes in length. Involvement and coping will be emphasized through active forms of music participation, including drum circles, unit playlist creation, song writing, jam sessions, and song discussion.
  Arms: Music Therapy

SUMMARY:
Workplace stress for healthcare workers is at an all-time high and the COVID-19 Pandemic magnified and amplified the impact of stress and burnout on health care workers, especially for frontline staff such as nurses. There are multiple external and individual factors that affect clinician well-being, and organizational factors are an important aspect to address when attempting to mitigate nurse burnout and improve well-being. This project seeks to expand two interventions that were piloted in the last few years since the Covid-19 Pandemic, validated to show improvement in staff well-being and decreased feelings of burnout following the interventions, and are easily implemented to benefit nurses and other multidisciplinary health care workers and students in both the inpatient and outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

- English-speaking employees or students at Penn State Health and College of Medicine.

Exclusion Criteria:

- Non-English speaking individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
The number of subjects who state preference for having long-term access to the intervention. | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree
The number of subjects who report improvement of subject's energy level needed to complete immediate job responsibilities. | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree
The number of subjects who report improvement of subject's understanding of what is needed in the moment to overcome challenges. | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree
The number of subjects who report improvement navigating challenging or difficult situations in the workplace | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree
The number of subjects who report improvement in expressing thoughts, questions and feelings with colleagues situations in the workplace. | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree
The number of subjects who report improvement in feeling less isolated at work. | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree

SECONDARY OUTCOMES:
The number of subjects reporting the intervention was well facilitated. | Survey data will be collected at the end of the intervention up to 30 minutes post intervention.
  This will be measured on a Likert scale where 0 is strongly disagree and 5 is strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: ERIC R MESSNER, PhD, Principal Investigator — Penn State University

IPD SHARING:
Plan to Share IPD: Undecided